CLINICAL TRIAL: NCT02235792
Title: Chronically-recorded Deep Brain Nuclei/Hippocampal High Frequency Oscillations (HFOs) as Biomarkers of Neurologic Disease.
Brief Title: High Frequency Oscillations in Neurologic Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bryan T. Klassen, M.D., Consultant Neurology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-002360
Record Dates: First submitted 2014-07-14; First posted 2014-09-10 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Parkinson; Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deep Brain Stimulation 37604 Activa PC+S (Experimental): All subjects will undergo DBS using the 37604 Activa PC+S device (single arm study).
  Interventions: Device: Activa PC+S

INTERVENTIONS:
Device: Activa PC+S — The model 37604 Activa PC+S system is a multiprogrammable device that both delivers electrical stimulation and records bioelectric data through one or two leads implanted in the brain.

SUMMARY:
This study is designed to evaluate the high-frequency range deep brain oscillations (HFO) as pathologic markers in patients undergoing deep brain stimulation for epilepsy or Parkinson disease. Newly developed technology allows for the chronic recording of these brain signals at the same time as clinical stimulation is occuring. We will learn both whether these HFO correlate with disease activity and whether the HFO change in response to ongoing stimulation (potentially giving insight into the underlying mechanism of action of DBS).

DETAILED DESCRIPTION:
This study is designed to evaluate the high-frequency range deep brain oscillations (HFO) as pathologic markers in patients undergoing deep brain stimulation for epilepsy or Parkinson disease. Newly developed technology allows for the chronic recording of these brain signals at the same time as clinical stimulation is occuring. We will learn both whether these HFO correlate with disease activity and whether the HFO change in response to ongoing stimulation (potentially giving insight into the underlying mechanism of action of DBS). Study participants will undergo DBS in the same way as is usually done but will receive this newer battery with ability to record brain signals.

ELIGIBILITY:
Inclusion criteria:

1. Medically-refractory neurologic disease amenable to therapy with deep brain stimulation including:

   1. Idiopathic Parkinson disease with motor fluctuation, dyskinesia, and/or medically refractory tremor despite optimal medical management by a movement disorders neurologist.

      OR
   2. Unilateral or bilateral mesial temporal lobe (hippocampal) epilepsy with complex partial, and/or secondarily generalized seizures, that is:

      * confirmed through a combination of interictal scalp EEG, ictal scalp EEG under video monitoring, ictal SPECT scanning, and/or invasive EEG monitoring
      * disabling seizure counts >2 per month documented over a 3 month period
      * refractory to at least three antiepileptic drugs given at clinically appropriate maintenance doses resulting in therapeutic plasma levels (in cases where such levels have been established for that particular drug. Drug failures because of side- effects will not be counted toward this total.
      * determined to have mesial temporal lobe epilepsy that is not amenable to resective surgery according to consensus opinion among epileptologists on our institution's multidisciplinary Epilepsy Surgery Committee
2. Mayo Clinic Deep Brain Stimulation Committee approval for bilateral deep brain stimulation therapy obtained on routine clinical grounds and without reference to this protocol.
3. Age 18 to 75.
4. Ability and willingness to provide informed consent and participate in the study protocol.

Exclusion criteria:

1. Diagnoses other than those included in #1 above.
2. Comorbid nonepileptic behavioral events or psychogenic movement disorder.
3. Medical contraindications to DBS surgery.
4. Psychiatric comorbidities not under stable medical therapy.
5. Neurodegenerative dementia (cognitive dysfunction resulting from frequent seizure activity will not be an exclusion criteria).
6. Implanted electronically active medical device with the potential to interfere with intracranial recordings (ex. pacemaker, automatic implantable cardioverter defibrillator (AICD), active vagal nerve stimulator).
7. Pregnancy; women of child-bearing potential will be required to commit to using an effective method of contraception during the entire duration of the trial. If a subject becomes pregnant despite these precautions, she will be required to report that to our center within two weeks at which point explantation of the experimental device would be an option.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-07; Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Degree of correlation of recorded neural signatures with disease severity as determined by regression analysis | 26 weeks post deep brain stimulator implantation
  Regression analysis will be performed using the measures of clinical disease severity as the independent variables and the various HFO measurement conditions/parameters as dependent variables.
  HFO parameters to be analyzed will include: 1) total power within each recorded band and 2) frequency distribution as defined by the ratio of power within the higher HFO frequency band versus the lower HFO frequency band.
  Clinical disease severity will be determined by: 1) Unified Parkinson's Disease Rating Scale (UPDRS III) score in each of the various conditions for Parkinson Disease (PD) subjects, 2) motor diaries linked with each visit for PD subjects, and 3) seizure counts from the 4 weeks of seizure diary preceding each visit for epilepsy subjects.
  (Note: UPDRS is a rating scale used to follow the longitudinal course of Parkinson's disease. Part III is a clinician-scored monitored motor evaluation.)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Klassen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Van Gompel JJ, Klassen BT, Worrell GA, Lee KH, Shin C, Zhao CZ, Brown DA, Goerss SJ, Kall BA, Stead M. Anterior nuclear deep brain stimulation guided by concordant hippocampal recording. Neurosurg Focus. 2015 Jun;38(6):E9. doi: 10.3171/2015.3.FOCUS1541. PMID 26030709
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials